CLINICAL TRIAL: NCT00775580
Title: Single Dose Two-Way Crossover Fasted Bioequivalence Study of Atenolol 100 mg Capsules in Healthy Volunteers
Brief Title: Bioequivalence Study of Atenolol 100mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-310
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence Atenolol Tablets
MeSH Terms: interventions — Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): atenolol 100 mg Capsules of Ranbaxy
  Interventions: Drug: Atenolol 100mg Tablets
- 2 (Active Comparator): Tenormin 100mg capsules
  Interventions: Drug: Atenolol 100mg Tablets

INTERVENTIONS:
Drug: Atenolol 100mg Tablets

SUMMARY:
The purpose of this study was to determine the bioequivalence of atenolol formulations after administration of single doses to normal healthy subjects under fasted conditions. These data were to be evaluated statistically to determine if the products meet bioequivalence criteria.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioequivalence study on atenolol comparing atenolol 100mg tablets of Ranbaxy with Tenormin 100mg capsules in healthy, adult, human, subjects under fasting conditions.

A total of 36 non-smoking subjects (26 men and 10 women) were included in this study, of which 35 finished the study according to the protocol,

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects at least 18 years of age.
2. Informed of the nature of the study and given written informed consent.
3. Have a body weight within 15% of the appropriate range as defined in the 1983 Metropolitan Life Company tables weighing at least 110 pounds.

Exclusion Criteria:

1. Hypersensitivity to Atenolol (Tenormin®) or related compounds such as propranolol (Inderal®).
2. Conditions that affect the absorption, metabolism or passage of drugs out of the body, e.g., sprue, celiac disease, Crohn's disease, colitis, liver, kidney or thyroid conditions.
3. Recent history (within one year) of mental illness, drug addiction, drug abuse or alcoholism.
4. Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
5. Received an investigational drug within the 4 weeks prior to study dosing.
6. Currently taking any prescription medication, except for oral contraceptives, within the 7 days prior to study dosing or over-the-counter medication within 3 days of study dosing. This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician. Any nonprescription medication consumption reported will be reviewed by the investigator(s) prior to dosing. At the discretion of the investigator(s), these volunteers may be enrolled if the medication is not anticipated to alter study integrity.
7. Regular smoking of more than 5 cigarettes daily or the daily use of nicotine-containing products beginning 3 months before study medication administration through the final evaluation.
8. If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the treatment periods. Females must use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral contraceptives/patches, progestin injection or implants, condom with spermacide, diaphragm with spermacide, IUD, vaginal spermicidal/hormonal suppository, surgical sterilization of themselves or their partner(s) or abstinence. Females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-05; Primary Completion 2005-05 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- aaiPharma, Inc. -AAI Clinic, Chapell Hill, North Carolina, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com.
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html